CLINICAL TRIAL: NCT05067361
Title: Effectiveness of Aerobic Exercises on the Stereotypic Behaviors and Task Performance of Autistic Children: A Randomized Clinical Trial
Brief Title: Effectiveness of Aerobic Exercises on the Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Amna Ayub PT, Physical Therapist, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TUF/DR/MSPP/173
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Physical therapy; Stereotypic behaviors; ASD; Repetitive behaviors; Aerobic exercises; Jogging; Ball exercises.
MeSH Terms: conditions — Autism Spectrum Disorder; Stereotypic Movement Disorder | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Procedure: Aerobic Exercise; Procedure: Ball Exercises
- Active control Group (Active Comparator)
  Interventions: Procedure: Ball Exercises

INTERVENTIONS:
Procedure: Aerobic Exercise — Jogging was performed for 20 minutes. Jogging was performed by experimental group for 3 weeks and 4 sessions per week.
  Arms: Experimental Group
Procedure: Ball Exercises — Ball exercises like stability ball roll, stability ball hug, stability ball catching, ball throwing and ball tapping exercises were for 10 minutes. Ball exercises was performed by both groups for 3 weeks and 4 times per week .

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder manifesting stereotypic behaviors and problem in communication and social interaction. Different physical therapy interventions like aerobics help to improve recurrent behaviors and task performance of autistic children. This study was focused to see the effect of jogging on the stereotypic behaviors and task performance of autistic children. A single blinded randomized study was conducted on 38 autistic children, randomly allocated to two groups, performing jogging and ball exercises. Repetitive Behavior Scale-revised(RBS-R) and Jebsen Hand Function Test (JHFT) was used for assessment. Exercise was performed for 3 weeks and 4 sessions per week.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed children of autism spectrum disorder (ASD) by experts
2. Have recognized stereotypic behaviors
3. Age 6 to 20 years
4. Independent to walk
5. Both genders
6. Parent and teachers willing to give consent

Exclusion Criteria:

1. Unable to understand commands
2. Have co-morbidities like schizophrenia or ADHD
3. Having respiratory or cardiovascular problems
4. Severe ASD
5. Lower limb injury and disability

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Repetitive behavior scale revised (RBS-R) | 3 weeks
  RBS-R was used to assess the stereotypic behaviors of autistic children. It is 43 items questionnaire that is placed under six subscales. The sub-scales are Stereotyped Behavior Subscale Self-Injurious Behavior Subscale Compulsive Behavior Subscale Ritualistic Behavior Subscale Sameness Behavior Subscale Restricted Behavior Subscale Each subscale has different characteristics, which are classified from 0 to 3 (behavior is severe). Moreover, each behavior is also rated that how much this behavior occurs, cause interruption in activity and how much a child become agitated when he was interrupted. Global score rating was used by calculating the scores of all the six subscales and total score was given in range of 1 to 100.

SECONDARY OUTCOMES:
Jebsen Hand Function Test (JHFT) | 3 weeks
  JHFT was used to evaluate the task performance of autistic children.JHFT has seven variants and time was recorded, in seconds, taken by children to complete these seven tasks. These seven tasks are writing, card turning, small common objects, simulated feeding, stacking, lifting large lightweight objects and lifting large heavy objects. These piece of work was first performed by the non-dominant hand then by the dominant hand and at the end time required during all the task was summed up in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sidra Majeed;PT, MSPP, Study Director — University of Faisalabad
Locations (1):
- University of Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No